CLINICAL TRIAL: NCT00393900
Title: Middle Ear Pressure Disregulation After Tympanostomy Tube Insertion
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Ellen M. Mandel, Associate Professor, University of Pittsburgh
Other Study IDs: #0605013; NIH 1P50DC007667
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Otitis Media With Effusion
Keywords: otitis media; tympanostomy tube; eustachian tube function; gas exchange; tympanostomy tubes
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal cells obtained for DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children with tympanostomy tubes for chronic OME

SUMMARY:
This study will determine if the investigators can use certain tests (eustachian tube function tests and gas exchange tests) to predict whether or not a child who had tubes surgically placed in their eardrum because of middle-ear disease will redevelop the disease again after the tubes quit working.

DETAILED DESCRIPTION:
This study will enroll children 3-6 years of age with tympanostomy tubes inserted for otitis media with effusion (OME)and measure middle ear gas demand, middle ear volume and eustachian tube function longitudinally between the time of tube insertion and extrusion/nonfunctioning. The data will be used to test the hypotheses that: gas transfer across the middle ear mucosa decreases in phase with resolution of middle ear inflammation and effusion; gas transfer across the middle ear mucosa is increased by an episode of otorrhea; eustachian tube function is unaffected by tympanostomy tube insertion, and measurement of eustachian tube function and trans-middle ear mucosa gas transfer predicts disease recurrence and presentation after tube extrusion/nonfunctioning. The results of these studies will be used to support or refute tested components of existing models of middle ear pressure-regulation and to develop test protocols for risk assignments with respect to disease recurrence in individual ears after tympanostomy tube extrusion/nonfunctioning.

ELIGIBILITY:
Inclusion Criteria:

* 3-6 years old
* History of chronic otitis media with effusion(OME)
* Scheduled or within 6 weeks of tube insertion
* OME at entry or surgery
* Generally good health

Exclusion Criteria:

* Cleft palate or other syndromes predisposing to OM
* History of recurrent acute otitis media only
* History of complications of OM or its treatment
* Unable to cooperate for testing

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 3-6 years old who underwent tympanostomy tube insertion for chronic otitis media with effusion within the 6 weeks prior to study enrollment
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
middle ear status | 12 months
  middle-ear status at 12 months after tympanostomy tube became non-functional

CONTACTS AND LOCATIONS:
Overall Officials: William J Doyle, PhD, Principal Investigator — Department of Otolaryngology, Children's Hospital of Pittsburgh; Ellen Mandel, MD, Study Director — University of Pittsburgh
Locations (1):
- ENT Department, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mandel EM, Swarts JD, Casselbrant ML, Tekely KK, Richert BC, Seroky JT, Doyle WJ. Eustachian tube function as a predictor of the recurrence of middle ear effusion in children. Laryngoscope. 2013 Sep;123(9):2285-90. doi: 10.1002/lary.24021. Epub 2013 Apr 10. PMID 23575552